CLINICAL TRIAL: NCT06557915
Title: Evaluation of Nasal Problems in Neonates and Infants Subjected to CPAP in Sohag University Hospitals
Brief Title: Nasal Problems in Neonates and Infants Subjected to CPAP
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abdelaal, Evaluation of nasal problems in neonates and infants subjected to CPAP in Sohag University hospitals, Sohag University
Other Study IDs: Soh-Med-24-07-05MS
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Continuous Positive Airway Pressure
Keywords: neonates; CPAP
MeSH Terms: interventions — Mass Screening

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neonates and Infants Subjected to CPAP: * Detection and Screening of different nasal complications of using CPAP in neonates and infants
  * reach a consensus about minimizing nasal problems of CPAP in neonates and infants
  Interventions: Procedure: screening

INTERVENTIONS:
Procedure: screening — screening and detection of nasal problems in Neonates and Infants Subjected to CPAP

SUMMARY:
The goal of this study is to Detect and Screen different nasal complications of using CPAP in neonates and infants and reach a consensus about minimizing nasal problems of CPAP in neonates and infants

DETAILED DESCRIPTION:
Continuous Positive Airway Pressure (CPAP) is a means of providing respiratory support to neonates with either upper airway obstruction or respiratory failure. Respiratory failure constitutes either failure of ventilation or failure of lung function.

Nasal CPAP can be delivered through various devices, of which a nasal mask and binasal prongs are the most commonly used. However, earlier studies have described the development of Pressure Injuries (PI) on the nasal skin caused by these nCPAP devices

Nasal complications of nasal CPAP vary from external nasal complications such as columellar hyperemia, columellar necrosis to intranasal complications such as intranasal ulceration, granulation, vestibular stenosis and intranasal synechiae

Aims of the Study:

* Detection and Screening of different nasal complications of using CPAP in neonates and infants
* reach a consensus about minimizing nasal problems of CPAP in neonates and infants

Patients and Methods:

* Type of the study: prospective study.
* Place of the study:

  * Pediatric department and its units (Neonatal intensive care unit (NICU), Pediatric intensive care unit (PICU), Critical care unit)
  * Otorhinolaryngology department In Sohag university hospitals (old and new)
* Study period: One year from date of acceptance of the protocol.
* Patient:

Neonates and infants subjected to CPAP and presented to ENT department for assessment of nasal condition

• Methods:

All cases will be subjected to:

1. Full medical history: Name, age, sex, date of birth
2. Indications and duration of CPAP
3. Complete Ear,nose and throat (ENT) examination including endoscopic examination

ELIGIBILITY:
Inclusion Criteria:

* Neonates and infants subjected to CPAP and presented to ENT department for assessment of nasal condition

Exclusion Criteria:

* Failure to obtain consent.
* Children above 1 year
* Adults

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All neonates (full and preterm), infants (less than 1 year) subjected to CPAP with different indications
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Detection of different nasal complications of using CPAP in neonates and infants | 1 week following using CPAP in neonates and infants
  the metric used is complete ENT examination of neonates and infants subjected to CPAP

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdelaal, Principal Investigator — faculty of medicine,sohag university
Locations (1):
- Faculty of Medicine, Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided